CLINICAL TRIAL: NCT05830448
Title: Evaluation of the Effect of Cognitive Behavioral Approach-Based Stress Coping Skills Training Program Performed by Tele-Nursing on Stress Perception, Resilience and Compassion Fatigue in Palliative Care Nurses
Brief Title: Evaluation of the Effect of Cognitive Behavioral Approach-Based Stress Coping Skills Training Program on Stress Perception, Resilience and Compassion Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ozge AYDOGAN ASIR, Principal İnvestigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OZGE AYDOGAN ASIR; OZLEM ORSAL (Other: EskişehirOU)
Record Dates: First submitted 2023-01-31; First posted 2023-04-26 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Stress Perception, Psychological Resilience, Compassion Fatigue
Keywords: palliative care nurses; Stress; Stress Perception; Ability to Cope with Stress; Psychological Resilience; Compassion Fatigue
MeSH Terms: conditions — Compassion Fatigue | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Experimental study with randomized pretest-posttest control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The nurses to be included in the study will be assigned to the intervention and control groups by simple randomization using the computer-assisted randomization application (www.randomizer.org). Determination of the intervention and control group will be drawn between set1 and set2. The ranking to be given to the participants (eg 1,2,3,….32) will be created by recording the number of participants when they approve to participate in the research (eg, the 10th person who accepts to participate will automatically be the 10th participant). No new applications will be accepted when the number of people to be included in the sample is reached. Participants in the study will not know which group they belong to. The researcher will contact the individual assigned to the control and intervention group according to the number given without knowing who the participant is. Blinding will be provided by Outcomes Assessor during data entry and statistics stages.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Experimental): CBD is a model that applies learning theories to assist people when they encounter difficulties and life problems that they cannot cope with in their daily lives. It focuses on the elements that affect emotions and behaviors, that is, the thought system. CBT is a process that involves changing the automatic thoughts and evaluations that occur when people are faced with negative situations with different thoughts that can create alternatives and restructuring these thoughts. The approach essentially argues that the way events are perceived and interpreted is more important than how they happen. Systematic errors in information processing, which cause people to perceive themselves, their environment and their future negatively, cause stress and symptoms of mental disorders. There are studies showing that cognitive behavioral therapy reduces stress levels and stress symptoms.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Mobile Mental Health Support System created by the Turkish Ministry of Health (Active Comparator): This system aims to protect and support the mental health of the health personnel of the Ministry of Health. It is a mobile application that allows video calls with a secure and official channel with voluntary adult and child-adolescent mental health and diseases specialists for himself and his children. Personnel who want to benefit from the said service will be able to access the service by downloading the Ministry of Health RUHSAD application to their mobile devices after searching for "Mental Health Support System" in the mobile application markets and following the instructions.
  Interventions: Behavioral: T.R. Mobile Mental Health Support System produced by the Ministry of Health

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The trial was planned to have a three-month announcement and an eight-week intervention period. Personal information form, Perceived Stress Scale, Coping with Stress Scale, Connor-Davidson Resilience Scale, Quality of Life Scale for Employees will be used in the pre-test phase of data collection. Participants meeting the inclusion criteria will be randomly assigned to the intervention and control groups. In order to support nurses in the intervention group to gain awareness of stress and anxiety and develop positive coping skills, 8 sessions of 40 minutes were planned, including interaction steps based on education and cognitive approach. As of the second week, homework will be given to individuals and they will be asked to submit these assignments to the researcher 2 days before the next interview. Participants who do not submit the assignments given in this study to the researcher on time will be excluded from the study even if they have completed the training.
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: T.R. Mobile Mental Health Support System produced by the Ministry of Health — No intervention will be applied to the individuals assigned to the control group by the researcher. Participants will be informed about the Mobile Mental Health Support System created by the Turkish Ministry of Health and will be directed to this application.
  Arms: Mobile Mental Health Support System created by the Turkish Ministry of Health

SUMMARY:
This research is an experimental study with a randomized pre-test-post-test control group to evaluate the effect of the cognitive behavioral approach-based stress coping skills training program carried out by tele-nursing on the palliative care nurses' perception of stress, resilience and compassion fatigue.

The main questions it aims to answer are:

Question 1. Will the cognitive behavioral approach-based stress coping skills training program to be carried out through tele-nursing have an effect on the increase in the stress coping score of the palliative care nurses in the intervention group? Question 2. Will the cognitive behavioral approach-based stress coping skills training program to be carried out through tele-nursing have an effect on the reduction of stress perception among palliative care nurses in the intervention group? Question 3. Will the cognitive behavioral approach-based stress coping skills training program to be carried out through tele-nursing have an impact on the increase in resilience of palliative care nurses in the intervention group? Question 4. Will the cognitive behavioral approach-based stress coping skills training program to be carried out through tele-nursing have an effect on the reduction of compassion fatigue in palliative care nurses in the intervention group? The research was planned as a randomized controlled experimental design with the required ethics committee and institution permissions, a three-month announcement and initiation period, and an eight-week intervention period. Data will be collected twice at baseline and after intervention (Week 9). Personal information form, Perceived Stress Scale, Coping with Stress Scale, Connor-Davidson Resilience Scale, Quality of Life Scale for Employees will be used in the pre-test phase of data collection. Participants meeting the inclusion criteria will be assigned to the intervention and control groups by randomization. In order to support nurses in the intervention group to gain awareness of stress and anxiety and develop positive coping skills with stress, a total of 8 sessions of 40 minutes are planned, including interaction steps based on education and cognitive approach. Individuals will be given homework from the second week and they will be asked to deliver these homeworks to the researcher 2 days before the next interview, and it is planned to send reminder messages from the WastApp group created. Participants who do not deliver the assignments given in this study to the researcher on time will be excluded from the research even if they participate in online training.

No intervention will be applied to individuals assigned to the control group. Participants will be informed about the Mobile Mental Health Support System created by the Turkish Ministry of Health and will be directed to this application.

It is planned to apply Perceived Stress Scale, Coping with Stress Scale, Connor-Davidson Resilience Scale, Quality of Life Scale for Employees at the 9th week for the application of post-tests.

ELIGIBILITY:
Inclusion criteria:

* Working as a nurse in designated hospitals in Eskişehir,
* To have been working in palliative care services for at least one month,
* Having active internet access and being able to actively use a computer/tablet or smart phone.
* Volunteering to participate in the research.

Exclusion Criteria:

* Working in hospitals located in other provinces of Turkey,
* Working in all units in hospitals except the palliative care service,
* Having any psychiatric diagnosis other than stress,
* Being currently receiving psychological counseling,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-10-12 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | 5 months
  The stress perception of the nurses working in the palliative care service will be evaluated. The minimum score that can be obtained from the perceived stress scale is 0, and the maximum score is 56. A higher score on this scale means a worse result.
Connor-Davidson Resilience Scale | 5 months
  The psychological resilience levels of the nurses working in the palliative care service will be evaluated. The minimum score that can be obtained from the Connor-Davidson Resilience scale is 0, and the maximum score is 100. A higher score on this scale means a better result.
Quality of Life Scale for Employees - Compassion Fatigue Sub-Dimension | 5 months
  Information about compassion fatigue of nurses working in palliative care service will be given. The minimum score that can be obtained from the Employee Quality of Life Scale - Compassion Fatigue Sub-Dimension is 0, and the maximum score is 50. A higher score on this scale means a worse result.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi Universty, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No